CLINICAL TRIAL: NCT00440492
Title: An Open-Label Study To Evaluate The Potential Pharmacokinetic Interaction Between PLA-695 And Methotrexate When Coadministered Orally To Adult Subjects With Rheumatoid Arthritis
Brief Title: Study To Evaluate The Pharmacokinetic Interaction Between PLA-695 And Methotrexate In Adults With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3175A3-104
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — PLA-695

INTERVENTIONS:
Drug: PLA-695

SUMMARY:
The purpose of this study is to determine if PLA-695 changes the blood concentrations of methotrexate when administered together.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential with rheumatoid arthritis (RA), aged 18 to 75 years
* RA disease onset after 16 years of age and has had the disease for at least 6 months
* Must be receiving a stable, well-tolerated oral dose of methotrexate (5 to 25 mg) taken once weekly for at least 3 months

Exclusion Criteria:

* Evidence of unstable clinically significant disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of PLA-695 on the blood concentrations of methotrexate when administered together.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (9):
- United States (6):
  - Los Angeles, California
  - Palo Alto, California
  - Lake Success, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Columbus, Ohio
- Canada (3):
  - Vancouver, British Columbia
  - Mississauga, Ontario
  - Montreal, Quebec